CLINICAL TRIAL: NCT02730286
Title: Factors Associated With Activity Limitations in Individuals With Rheumatoid Arthritis
Brief Title: Activity Limitations in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Júnia Amorim Andrade, PHD Júnia Amorim Andrade, Federal University of Minas Gerais
Other Study IDs: MS ID#: AJOT/2015/017467
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Rheumatoid Arthritis
Keywords: human activity; International Classification of Functioning
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Observation

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational study — application of several standard instruments in patients with rheumatoid arthritis

SUMMARY:
Objective: To evaluate what factors contribute to activity limitations in subjects with rheumatoid arthritis considering the International Classification of Functioning, Disability and Health model.

Methods: A cross-sectional study on 81 individuals with rheumatoid arthritis (RA) using instruments to measure five constructs of the component activities.

DETAILED DESCRIPTION:
The investigators used the ICF model to analyze factors reported to be associated with functioning and disability in individuals with RA, including dexterity fatigue, stiffness , pinch, handgrip, strength, range of motion (ROM) deficit, deformities , mental health, vitality, and pain .

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years,
* Clinical diagnosis rheumatic arthritis
* Mental competence by the Mini-Mental State Examination

Exclusion Criteria:-

* Had undergone upper limb surgery,
* Had an uncorrected visual deficit that could compromise functionality

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For this cross-sectional study, 81 patients treated between June 2009 and August 2010 in Clinics Hospital, at the Universidade Federal de Minas Gerais (UFMG) in Brazil were recruited by convenience sampling
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Model 1- Test d´Evaluation dês Membres Supérieurs de Personnes Agées, - TEMPA rheumatoid arthritis | up to thirty minutes
  The TEMPA is assessing the performance of the upper extremities and consists of eight standardized tasks. Scoring of the task analysis dimension ranges from zero to 150 (a score of zero indicates no disability). The TEMPA is scored according to the time required (in seconds) to complete each task; the higher the score, the greater the disability
Model 2- Sequential Occupational Dexterity Assessment (SODA) | up to thirty minutes
  The SODA in patient population with RA score ranges from zero to 108 across these 12 tasks, has been validated for RA patients
Model 3 and 4- SF-36=Short form health survey-36 | up to thirty minutes
  The SF-36 has eight scales and a final score ranging from zero to 100 for each of the eight dimensions (a score of 100 represents the best state of health). The Brazilian Portuguese version of the SF-36 in patient population with RA has been demonstrated to be a reproducible and valid.
Model 5 - AIMS=Arthritis impact measurement scale | up to thirty minutes
  The score ranges from zero to 10 (a score of 10 indicates the worst state of health) in patient population with RA. The Portuguese version of AIMS2 has been shown to be satisfactory

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andrade JA, Brandao MB, Pinto MR, Lanna CC. Factors Associated With Activity Limitations in People With Rheumatoid Arthritis. Am J Occup Ther. 2016 Jul-Aug;70(4):7004290030p1-7. doi: 10.5014/ajot.2016.017467. PMID 27294995